CLINICAL TRIAL: NCT03517670
Title: Safety of Intravenous Milrinone for the Treatment of Subarachnoid Hemorrhage-induced Vasospasm
Acronym: MilriSpasm
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC17_0451
Record Dates: First submitted 2018-04-23; First posted 2018-05-07 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-03

CONDITIONS: Cerebral Vasospasm; Subarachnoid Hemorrhage
Keywords: Cerebral vasospasm; Subarachnoid hemorrhage; Milrinone; Hemodynamic tolerance
MeSH Terms: conditions — Vasospasm, Intracranial; Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Rhythmic tolerance — Rhythmic intolerance is defined by the occurrence of arrhythmia prompting the initiation of an antiarrhythmic medication and the need to decrease or even to stop the infusion of milrinone
Other: Hematological tolerance — Hematological tolerance will be considered good if milrinone infusion was not interrupted owing to the occurrence of thrombocytopenia
Other: Milrinone efficiency on cerebral vasospasm — It will be assessed using ultrasound measurements of middle cerebral arteries velocities. A decrease of at least 20% of the mean velocity or of the Lindegaard index will be considered as a significant positive effect of the treatment (including milrinone).
Other: Milrinone efficiency using the modified Rankin scale — Scored as follows: 0 = No symptoms, 1 = No significant disability. Able to perform all usual activities, despite certain symptoms, 2= Slight disability. Able to take care of his own affairs without assistance, but unable to carry out all previous activities, 3 = Moderate disability. Requires some help, but able to walk unassisted, 4 = Moderate severe disability. Unable to meet their own physical needs without help and unable to walk without help, 5 Severe disability. Needs constant care and attention, bedridden, incontinent, 6 = Death.

SUMMARY:
The aim of this study is to evaluate the tolerance of intravenous milrinone combined to the current standard treatment for cerebral vasospasm following subarachnoid hemorrhage. Assessment of IV milrinone safety in this setting is mandatory before the conduction of a large study assessing its effectiveness.

DETAILED DESCRIPTION:
The aim of this prospective observational study is to evaluate the hemodynamic tolerance of intravenous milrinone for the treatment of arterial vasospasm following subarachnoid hemorrhage. Intravenous milrinone is part of our standard care protocol for the management of cerebral vasospasm in association with nimodipine (intravenous or enteral route) and high arterial blood pressure (mean arterial pressure of 100-120 mmHg, spontaneously or induced by volume expansion and norepinephrine). All patients of our ICU who were diagnosed with cerebral arterial vasospasm during the few days following a subarachnoid hemorrhage will be included.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18 years
* Hospitalized in our intensive care unit
* Subarachnoid hemorrhage proven on CT angiogram
* Cerebral vasospasm proven on CT angiogram

Exclusion Criteria:

* Pregnant women
* Minor
* Major under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary Purpose: Treatment Study Phase: NA Intervention Model: Single group Number of Arms: 1 Masking: Open label Allocation: NA Study Endpoint Classification: Safety Enrollment: 60 participants
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-08-31 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Hemodynamic tolerance during treatment: defined by a stable mean blood pressure of 100-120 | At 6 months.
  A good hemodynamic tolerance is defined by a stable mean blood pressure of 100-120 mmHg without neither the need to decrease milrinone infusion rate below 0.5 g.kg-1.min-1 nor the need to increase norepinephrine above 1g.kg-1.min-1 Safety Issue: No

SECONDARY OUTCOMES:
Rhythmic tolerance: defined by the occurrence of arrhythmia prompting the initiation of | Rhythmic tolerance will be assessed for the duration of treatment, which will be on average one month.Heart rate and rhythm will be measured continuously, but assessed for fluctuation outside the reference range daily (during the length of treatment).
  Rhythmic intolerance is defined by the occurrence of arrhythmia prompting the initiation of an antiarrhythmic medication and the need to decrease or even to stop the infusion of milrinone Safety Issue: No
Hematological tolerance: will be considered good if milrinone infusion was not interrupted | Hematological tolerance will be assessed daily through measuring platelet count for the duration of treatment.
  Hematological tolerance will be considered good if milrinone infusion was not interrupted owing to the occurrence of thrombocytopenia Safety Issue: No
Milrinone efficiency on cerebral vasospasm | Milrinone efficiency on cerebral vasospasm will be assessed for the duration of treatment, which will be on average one month. Mean velocity and the lindegard index will be initially measured at 0, 2, 12 and 24 hours; and subsequently daily.
  It will be assessed using ultrasound measurements of middle cerebral arteries velocities. A decrease of at least 20% of the mean velocity or of the Lindegaard index will be considered as a significant positive effect of the treatment (including milrinone).
  Safety Issue: No
Milrinone efficiency on patient-centered neurological outcome using the modified Rankin scale | At 6 months.
  Scored as follows: 0 = No symptoms, 1 = No significant disability. Able to perform all usual activities, despite certain symptoms, 2= Slight disability. Able to take care of his own affairs without assistance, but unable to carry out all previous activities, 3 = Moderate disability. Requires some help, but able to walk unassisted, 4 = Moderate severe disability. Unable to meet their own physical needs without help and unable to walk without help, 5 Severe disability. Needs constant care and attention, bedridden, incontinent, 6 = Death.
  Safety Issue: No

CONTACTS AND LOCATIONS:
Overall Officials: Julien CADIET, PH, Principal Investigator — Nantes University Hospital
Locations (1):
- CHU Nantes, Nantes, France